## Study Protocol

#### Official title:

The Relationship Between CES1 Genotype and Methylphenidate Response in Children With ADHD - INDICES Work Package 6

Date of approval from human subject protection review board:

22<sup>nd</sup> March 2012

#### Short summary:

This is a prospective observational study of a cohort of children diagnosed with Attention Deficit Hyperactive Disorder (ADHD) and followed with weekly assessments during the first 12 weeks of Methylphenidate (MPH) treatment. The study was extended to include a three-year follow-up which is described in the additional protocol "Predictors of long-term outcome in a clinical cohort of children with attention-deficit hyperactivity disorder (ADHD)".

| Table of content | Pages |
|---------------------------------------------|--------------|
| Original protocol – 12 week study | <u>3</u> -12 |
| Additional protocol – three year follow-up | 13-27 |
| Summary of amendments of the study protocol | 28 |

# The relationship between CES1 genotype and methylphenidate response in children with ADHD – INDICES workpackage 6 Protocol version 3

Tine Houmann<sup>1</sup>, Pia Jeppesen<sup>1</sup>, Kerstin von Plessen<sup>2</sup>, Anne-Katrine Pagsberg<sup>2</sup>, Kristine Kaalund Jørgensen<sup>1</sup>, Jan Buitelaar <sup>3</sup> Henrik Berg Rasmussen<sup>4</sup>

<sup>1</sup>Child and Adolescent Psychiatric Center Glostrup, University of Copenhagen, Denmark, <sup>2</sup>Child and Adolescent Psychiatric Center Bispebjerg, University of Copenhagen, Denmark, <sup>3</sup> Radboud University Nijmegen Medical Center, <sup>4</sup>Research Institute of Biological Psychiatry, Mental Health Centre Sct. Hans, Copenhagen University Hospitals, Denmark

INDICES: (Individualised drug therapy based on pharmacogenomics: Focus on carboxylesterasel) **SUMMARY.** 

We wish to examine the relationship of Carboxylesterase 1(CES1) genotype with the response to Methylphenidate (MPH) in children with attention deficit hyperactivity disorder (ADHD). This will allow us to develop guidelines for individualized CES1 genotype-based MPH treatment in patients with ADHD.

The INDICES project combines pharmacology, genetics and metabolomics with clinical psychiatry and cardiology. It consists of 7 workpackages with focus upon carboxylesterase 1 (CES1), an enzyme with a major role in the metabolism of a variety of essential drugs including methylphenidate (MPH) and trandolapril (TA) for treatment of ADHD and cardiovascular disease (CVD), respectively.

The overall aim is to develop and implement guidelines for individualized treatments with MPH and TA and obtain a better drug response and reduce the risk of adverse reactions.

#### **Background (Workpackage 6):**

MPH is first-line treatment for ADHD, which affects 3-5% of children and adolescents. In most cases it persists into adulthood<sup>1</sup>. In Denmark the consumption of MPH has increased by a factor of 10 during the last 10 years<sup>2</sup>

Comorbidity is common, affecting more than 80% of patients with ADHD.

15- 20 % of patients treated with MPH are nonresponders. Adverse reactions are common, but few studies have had adverse reactions as their primary focus<sup>3,4</sup>. Decreased appetite is closely linked to stimulant treatment, and sleep problems occurs in approximately 70% in the initial stages of treatment. Increased blood pressure and heart rate, associated with stimulant treatment, affects a minority of treated individuals (5%). Potentially more serious cardiovascular events, however, seem to appear in stimulant treated children, with a risk, similar to the background population <sup>5</sup>. Discontinuation of treatment because of adverse reactions occurs in 2-10% <sup>4</sup>. Overall, adverse reactions in MPH treatment seem to be linked to individual underlying mechanisms, possibly related to pharmacokinetics and pharmacogenomics. Guidelines for treatment with MPH emphasize the need for individually tailored medication dosage, and further research into pharmacogenetics, but the clinical use of these tools is still highly variable <sup>3,6,7</sup> Several studies have found evidence for genetic variations in MPH response, especially variations in the dopamine transporter and dopamine D4 receptor. Variations in candidate genes, predict differences in ADHD treatment response and side effects of immediate release MPH <sup>8-10</sup>

Carboxylesterase 1(CES1) is a key enzyme in the metabolism of MPH, various other drugs, and endogenous lipids. Clinical and preclinical studies indicate that polymorphisms in the CES1 gene are responsible for individual variations in MPH treatment response and drug-drug interactions <sup>11-13</sup>. Recent data from a collaborative study supported by the European Commission (EU-FP7) have revealed duplication of the CES1 gene at frequencies of approximately 0.20 in Europe (Henrik Berg Rasmussen, unpublished). Gene duplication may give rise to increased rate of metabolism of CES1 dependent drugs.

#### **Hypotheses:**

Our main hypotheses: Individuals with a gene variant of CES1 resulting in rapid metabolic breakdown of MPH will experience less therapeutic effect and thus need higher dosages. Individuals with a gene variant of CES 1 resulting in slow metabolizing of MPH will experience a better therapeutic effect and thus need lower dosages.

Our exploratory hypotheses: Dose-related side effects in MPH treatment will be associated with the metabolic rate of MPH breakdown, in line with its therapeutic effect.

#### Aims:

We aim to examine the influence of the CES1 genotype in children with ADHD on the effectiveness and the pharmacokinetics of MPH. Moreover, we aim to develop guidelines for individualised MPH therapy, based on CES1genotype by combining the results from INDICES Workpackage 2, a pharmacokinetic study of the correlation of CES1 genotype and copy number, with the pharmacokinetics of trandolapril and methylphenidate..

Implementation of guidelines for individualized pharmacotherapy will improve treatment efficacy and safety in this group of children.

#### **Studypopulation:**

200 drugnaïve children diagnosed with ADHD according to DSM-IV criteria in the age 7-12 years will be recruited from the three Child- and Adolescent Psychiatric Centers in the Capital Region of Copenhagen. To allow for a naturalistic setting, and because more than 80% of children and adolescents with ADHD have a comorbid psychiatric condition, we will only exclude patients with an IQ < 70, current serious medical or psychiatric illness (e.g. schizophrenia, bipolar disorder, untreated epilepsy, heart failure).

#### **Inclusion criteria:**

Age: 7-12 years (both inclusive)

Both sexes

DSM-IVADHD diagnosis (any subtype)

Clinical indication for methylphenidate treatment, based on national guidelines, confirmed by an ADHD-RS score +1.5 SD above mean adjusted for age and sex

Drug naïve to ADHD medication (Methylphenidate, Dexamphetamine, Atomoxetine)

Written informed consent by parents holding custody, and the child, to participate in the study

#### **Exclusion criteria:**

Medical conditions that contraindicate treatment with MPH: Cardiovascular or cerebrovascular disease, hyperthyroidism, phaeocromocytoma, glaucoma.

Psychiatric conditions that contraindicate treatment with MPH: Mania, psychosis, former severe depression, bipolar disorder not well controlled, suicidal conduct, anorexia nervosa

Diagnosis of mental retardation (IQ  $\leq$  70)

Any ADHD medication ever (Methylphenidate, Dexamphetamine, Atomoxetine)

Current treatment with another CES1 related drug (Tamiflu, Trandolapril)

Current treatment with antipsychotics

Treatment with irreversible MAO inhibitors within the last 14 days before treatment start

#### **Methods:**

The psychometric instruments used in this study, for diagnostic assessment, are standard procedures for children in the age group, referred with a possible diagnosis of ADHD, in the Capital Region of Copenhagen. The staffs (Child- and adolescent psychiatrists and psychologists) who are conducting the assessments at the three study sites have all been trained in the psychometric instruments used in this study. We will measure interrater-reliability (by using kappa) for the K-SADS interviews. The INDICES workpackage 6 study group includes a local child and adolescent psychiatrist, who is the responsible researcher on each of the three study sites.

#### **Diagnostic assessment:**

All children referred to the three Centers of Child and Adolescent Psychiatry in the Capital Region of Copenhagen, with a possible diagnosis of ADHD, are assessed by the following procedures: The CBCL<sup>14</sup> (web-based questionnaires)

K-SADS interview<sup>15</sup>

Clinical assessment and diagnosis of ADHD according to Danish national guidelines, including history of development, symptoms and sociodemographics, clinical observation of symptoms, cognitive test and standard physical examination

ADHD diagnosis confirmed by K-SADS

Comorbidity diagnosed with K-SADS.

Possible cases, based on age and ADHD diagnosis, are evaluated by the local responsible researcher for inclusion in the study, and if relevant, contacted for permission and written informed consent by parent(s) holding custody, and the child, to participate in the study

#### Baseline ratings and measures on patients meeting inclusion criteria:

ADHD-RS <sup>16</sup> rated by parent

ADHD-RS rated by teacher

Investigator rated ADHD-DSM-IV-RS <sup>17</sup>

CGI- Severity scale <sup>18</sup>

Connors CPT<sup>19</sup> or TOVA<sup>20</sup>(to be finally decided)

Adverse reactions-Rating Scale <sup>21</sup>

ASK-ME parent rated questionnaire, attitude scale (7 questions) <sup>22</sup>

Body weight and height

Blood pressure and pulse

#### **DNA samples:**

A sample of saliva

Patients included in the study enter a twelve week study period with dose escalation of methylphenidate, weekly telephone ratings and monthly clinical assessments of effect and adverse reactions to MPH treatment. Weekly telephone ratings are done by the PhD. student, and the following decision on pursuing further dose escalation is made in cooperation with the

child's regular psychiatrist at the study site. Monthly clinical assessments and decisions on dose escalation are done by the child's regular psychiatrist.

#### Weekly assessment and ratings:

(not made in week 4, 8 and 12)

By telephone: ADHD-DSM-IV-RS and Adverse Reaction-Rating Scale .

Weekly decision on pursuing further dose escalation based on the above ratings

#### **Clinical assessment:**

Every four weeks:

Measurement of blood pressure, pulse, weight and height

ADHD-DSM-IV-RS

Parent rated ADHD-RS

Adverse reactions-Rating Scale

#### Supplementary rating and test at week 8:

Teacher rated ADHD-RS

Blood test to measure serum concentration of Ritalin acid, and DNA

#### Outcome ratings after twelve weeks:

Investigator rated ADHD-DSM-IV-RS (primary outcome measure)

CGI-Severity (secondary outcome measure)

CGI-Improvement (secondary outcome measure)

CGI-Efficacy (secondary outcome measure)

Connors CPT or TOVA(secondary outcome measure)

Parent rated ADHD-RS (secondary outcome measure)

Teacher rated ADHD-RS (secondary outcome measure)

Adverse reactions-Rating Scale (secondary outcome measure)

#### **Outcome measures:**

Investigator rated ADHD-DSM-IV-RS score

Parent rated ADHD-RS score

Teacher rated ADHD-RS score

CGI-I

CGI-S

CGI-E

Connors or TOVA

MPH dose required for "Borderline normalisation" on ADHD-DSM-IV-RS: T-score 60-70

MPH dose required for normalisation on ADHD-DSM-IV-RS: T-score < 60

Occurrence (no. of weeks from treatment initiation) and type of adverse reactions

MPH dose at occurrence of adverse reaction

MPH dose at discontinuation, if that is necessary, because of adverse drug reactions or

Treatment failure (no effect of MPH on ADHD core symptoms)

Serum concentration of Ritalin acid at week 8

Body weight, height, blood pressure and pulse

#### **Dose escalation:**

MPH is initiated at a low dose: 5mg. MPH-IR three times daily (TID), and escalated weekly with 0 - 2,5 - 5mg MPH-IR TID. Maximum dose is 2mg/kg/day. MPH dose morning, midday and afternoon can be individually escalated, based on effect and adverse reactions. Decisions on dose escalation will be based on a clinical decision manual, elaborated for the study. Individual deviations in dose escalation are noted in the CRF and case records.

Dose escalation is continued on a weekly basis until one of the following:

- Normalisation on ADHD-RS defined as T-score < 60
- Borderline normalisation on ADHD-RS, if normalisation is not obtainable, defined as T-score 60-70
- Cessation of dose escalation because of adverse reactions
- Discontinuation of MPH because of either intolerable adverse reactions, or no effect of MPH on ADHD core symptoms.

On basis of this, we exploratively will categorize patients as

- 1) Clinically normal reponders
- 2) Clinically slow responders
- 3) Clinically rapid responders

#### **Results:**

We plan to use multivariate regression models with the change in symptom severity, measured with the ADHD-DSM-IV rating scale score as the dependent measure, whereas CES1genotype, weight adjusted MPH dosage (mg/kg/day), age, gender, occurrence of adverse reactions and ADHD subtype will serve as predictors.

We will repeat the analysis with CGI-I as the dependent measure.

This will allow us to assess whether MPH is less effective in subjects with CES1 gene variants, that are known to have a rapid metabolic breakdown of MPH, whether higher dosages of MPH, necessary to adapt to the genetic differences in these subjects, are associated with more side effects, whether subjects with CES1 gene variants that are known to have a slow metabolic breakdown of MPH, need lower dosages of MPH than expected, to have effect on ADHD core symptoms, and whether lower dosages of MPH, necessary to adapt to the genetic differences in these subjects, are associated with less side effects.

By combining our results with data from the pharmacokinetic work-package in the INDICES study, we will develop guidelines for individualised therapy of ADHD with MPH

#### **Ethics**

The clinical work package 6 focused on ADHD is covered by existing permissions from the local committees on scientific ethics (De Videnskabsetiske Komiteer for Region Hovedstaden) and the Danish Data Protection Agency (Datatilsynet). Those permissions allow the collection and examination of data as well as biological samples from psychiatric patients with ages below 18 years, for research purposes, including genetic research projects. Journal number: H-B-2009-026

#### Participating centres and collaborators:

Child and Adolescent psychiatric Center Glostrup, Copenhagen University Hospitals:

Tine Houmann (TH), Senior Consultant, Associate Professor, Pia Jeppesen (PJ), PhD, Post Doc,

Senior consultant, Associate Professor, Kristine Kaalund-Jørgensen (KKJ) MD

Child and Adolescent psychiatric Center Bispebjerg, Copenhagen University Hospitals:

Kerstin von Plessen (KP), PhD, Senior Consultant, Professor, Katrine Pagsberg (KP), PhD, Senior consultant, Associate Professor

Child and Adolescent psychiatric Center Hillerød, Copenhagen University Hospitals:

Jørgen Dyrborg (JD) Senior Consultant, Maj-Britt Lauritsen (MBL) MD

Radboud University Nijmegen Medical Center:

Jan K. Buitelaar (JB) Professor

Research Institute of Biological Psychiatry, Psychiatry Center Sct. Hans, Copenhagen University Hospitals:

Henrik Berg Rasmussen (HBR) PhD, Post doc

#### Milestones

2012: Month 1-2: planning and introduction

2012: Month 3-12: recruitment of 100 patients who will complete a 3-month study period of drugescalation

2013: Month 13-24: recruitment of 100 additional patients who will complete a 3-month study period corresponding to a total of 200

2014: Month 25-29: Finalization of entire clinical study. Data analysis. Preparation and submission of two manuscripts.

2014: Month 30-36: study visit at University of Nijmegen

2015: Month 37-39: Statistical treatment of data and elaboration of manuscripts. Advices for improved stimulant therapy developed

2015: Month 40-42: Preparation of PhD thesis. (Month 29-42: preparation of PhD thesis )

#### **Economy:**

The funding of this Research Project consists of a grant to the Parties from the Danish Strategic Research Council, and self financing.

WP6 DSF grant:

Scientific/academic salaries, 1 PhD student in 42 months: 1.650.000 Dkr.
Operating expenses in 42 months: 380.000 Dkr.
Overheads 3.1% 62.930 Dkr

Total DSF grant: 2.092.930 Dkr

WP6 Self-financing, Child and adolescent psychiatric center Glostrup:

Scientific/academic salaries, 42 months:

Technical/administrative salaries, 42 months:

Overheads 3,1%

288.000 Dkr.
90.000 Dkr.
11.718 Dkr.

Total self-financing: 389.718 Dkr.



#### **Outcome ratings:**

Investigator rated ADHD-DSM-IV-RS, CGI-I, CGI-S, CGI-E, parent rated ADHD-RS, teacher rated ADHD-RS, Connors-CPT/TOVA, Adverse reactions –RS

#### Reference List

(1) Pliszka S, AACAP work group.

Practice parameter for the assessment and treatment of children and adolescents with attention-deficit/hyperkinetic disorder.

2007

J Am Acad Child Adolesc Psychiatry 2007;4:894-921.

- (2) Danish Medicine Agency. MedStat. www laegemiddelstyrelsen dk, 2011Available from: URL: www.laegemiddelstyrelsen.dk,
- (3) Graham J, Banaschewski T, Buitelaar J, Coghill D, Danckaerts M, Dittmann RW, et al. European guidelines on managing adverse effects of medication for ADHD. 2011

Eur Child Adolesc Psychiatry 2011;20(1):17-37.

(4) Graham J, Coghill D.

Adverse effects of pharmacotherapies for attention-deficit hyperactivity disorder: epidemiology, prevention and management.

2008

CNS Drugs 2008;22(3):213-37.

(5) Hammerness PG, Perrin JM, Shelley-Abrahamson R, Wilens TE.

Cardiovascular risk of stimulant treatment in pediatric attention-deficit/hyperactivity disorder: update and clinical recommendations.

2011

J Am Acad Child Adolesc Psychiatry 2011;50(10):978-90.

(6) Pliszka S, AACAP work group.

Practice parameter for the assessment and treatment of children and adolescents with attention-deficit/hyperkinetic disorder.

2007

J Am Acad Child Adolesc Psychiatry 2007;4:894-921.

(7) Powell SG, Thomsen PH, Frydenberg M, Rasmussen H.

Long-term treatment of ADHD with stimulants: a large observational study of real-life patients.

2011

J Atten Disord 2011;15(6):439-51.

(8) Froehlich TE, McGough JJ, Stein MA.

Progress and promise of attention-deficit hyperactivity disorder pharmacogenetics. 2010

CNS Drugs 2010;24(2):99-117.

(9) Froehlich TE, Epstein JN, Nick TG, Melguizo Castro MS, Stein MA, Brinkman WB, et al. Pharmacogenetic predictors of methylphenidate dose-response in attention-

deficit/hyperactivity disorder.

2011

J Am Acad Child Adolesc Psychiatry 2011;50(11):1129-39.

(10) McGough JJ, McCracken JT, Loo SK, Manganiello M, Leung MC, Tietjens JR, et al. A candidate gene analysis of methylphenidate response in attention-deficit/hyperactivity disorder.

2009

J Am Acad Child Adolesc Psychiatry 2009;48(12):1155-64.

(11) Nemoda Z, Angyal N, Tarnok Z, Gadoros J, Sasvari-Szekely M. Carboxylesterase 1 gene polymorphism and methylphenidate response in ADHD. 2009

Neuropharmacology 2009;57(7-8):731-3.

(12) Zhu HJ, Appel DI, Peterson YK, Wang Z, Markowitz JS.

Identification of selected therapeutic agents as inhibitors of carboxylesterase 1: potential sources of metabolic drug interactions.

2010

Toxicology 2010;270(2-3):59-65.

(13) Xie S, Borazjani A, Hatfield MJ, Edwards CC, Potter PM, Ross MK. Inactivation of Lipid Glyceryl Ester Metabolism in Human THP1 Monocytes/Macrophages by Activated Organophosphorus Insecticides: Role of Carboxylesterases 1 and 2.

2010

Chem Res Toxicol 2010.

- (14) Achenbach T.M. Manual for the child Behavior Checklist/4-18 and 1991 Profile. Burlington VT: University of Vermont Department of Psychiatry; 1991.
- (15) Ambrosini PJ.

Historical development and present status of the schedule for affective disorders and schizophrenia for school-age children (K-SADS).

2000

J Am Acad Child Adolesc Psychiatry 2000;39(1):49-58.

- (16) DuPaul G, Power T, McGoey K, Ikeda M, Anastopoulos A. AD/HD Rating Scale IV: Checklists, norms, and clinical interpretation. New York: Guilford; 1998.
- (17) Zhang S, Faries DE, Vowles M, Michelson D.

ADHD Rating Scale IV: psychometric properties from a multinational study as a clinician-administered instrument.

2005

Int J Methods Psychiatr Res 2005;14(4):186-201.

(18) Berk M, Ng F, Dodd S, Callaly T, Campbell S, Bernardo M, et al.

The validity of the CGI severity and improvement scales as measures of clinical effectiveness suitable for routine clinical use.

J Eval Clin Pract 2008;14(6):979-83.

(19) Conners CK, Epstein JN, Angold A, Klaric J.

Continuous performance test performance in a normative epidemiological sample. 2003

J Abnorm Child Psychol 2003;31(5):555-62.

(20) Schatz AM, Ballantyne AO, Trauner DA.

Sensitivity and specificity of a computerized test of attention in the diagnosis of Attention-Deficit/Hyperactivity Disorder.

2001

Assessment 2001;8(4):357-65.

(21) Barkley RA, McMurray MB, Edelbrock CS, Robbins K.

Side effects of methylphenidate in children with attention deficit hyperactivity disorder: a systemic, placebo-controlled evaluation.

1990

Pediatrics 1990;86(2):184-92.

(22) Dosreis S, Zito JM, Safer DJ, Soeken KL, Mitchell JW, Jr., Ellwood LC.

Parental perceptions and satisfaction with stimulant medication for attention-deficit hyperactivity disorder.

2003

J Dev Behav Pediatr 2003;24(3):155-62.

# Predictors of long-term outcome in a clinical cohort of children with attention-deficit hyperactivity disorder (ADHD)

#### Tine Houmann

Senior consultant, Child and Adolescent Mental Health Center, Mental Health Services - Capital Region of Denmark, Department of Clinical Medicine, Faculty of Health Sciences, Copenhagen University

Attention-deficit hyperactivity disorder (ADHD) is a common developmental disorder that arises during childhood and involves difficulties in the acquisition and execution of specific intellectual, motor, or social functions. The course of severity and impairment in ADHD, have great individual variations and fluctuations over time, and has a chronic course in half of the affected individuals. Psychiatric comorbidity is common with prevalence rates between 50-80, but also, somatic comorbidity is reported with increased odds ratios compared to control groups, and ADHD is associated with significantly increased mortality rates due to especially accidents, also when controlled for conduct- and substance use disorders. Long-term cohort and register studies indicate that ADHD is associated with problems in the domains of education, employment status, suicidal behavior and risk behavior including accidents, substance use disorder and criminality. Studies of childhood predictors for adolescent and adult outcome in ADHD have identified severity of ADHD symptoms, psychiatric comorbidity, especially conduct disorder and major depressive disorder, female gender, IQ, low family income, and stressfull life events to predict a poorer outcome. Experience of poor treatment effect, side effects, and reluctance or forgetfulness in relation to medication have often been reported as reasons for discontinuation of ADHD medication<sup>39,45</sup>. Thus identification of predictors for successful treatment could aid in the decision of which treatment should be offered the individual patient with ADHD, in order to improve adherence and outcome. In studies of antipsychotics, early onset of antipsychotic effect, is shown to predict later clinical treatment response in psychotic disorders, also in children and adolescents(Stentebjerg-Olesen, Jeppesen et al. 2013). To our knowledge no studies have investigated time to treatment effect as a predictor for outcome in childhood ADHD.

The project makes use of systematically and prospectively collected data from a representative, consecutively recruited clinical cohort of 200 children, recently diagnosed with ADHD, who were closely monitored under standardized conditions during the first 12 weeks of Methylphenidate (MPH) treatment. We will use the existing prospective clinical data in this cohort and combine those with information's concerning risk- and psychosocial factors derived from parental reports and the Danish registries. Finally, we will follow the cohort after three years with respect to ADHD symptoms and impairment in daily life functioning. The findings, based on a systematic analysis of these associations, may aid the development of an evidence-based and individualized program for initiation and monitoring of drug- and psychosocial treatment in childhood ADHD with the main objective to improve the long-term prognosis of the disorder in the children.

#### **Objectives**

The primary aim of this study is to investigate if time to MPH treatment response is a predictor for the long-term symptomatic and functional outcome in a clinical cohort of children with ADHD. We hypothesized that response to MPH treatment after three weeks, during a 12 weeks treatment trial, independently of baseline level of symptoms, other child and family characteristics, and MPH response after 12 weeks, can

predict the outcome after three years. The secondary aim is to describe the course of ADHD symptoms and level of functional impairment three years after initiation of ADHD treatment.

#### The following hypotheses will be tested:

- Early treatment response defined as ≥ 20% reduction in clinician rated ADHD symptoms between baseline and week three, will predict symptom severity and level of functioning in daily life activities three years after baseline, independently of baseline level of symptoms, and other child and family characteristics
- Treatment response after 12 weeks, defined as ≥ 40% reduction in clinician rated ADHD symptoms between baseline and week 12, will predict symptom severity and level of functioning in daily life activities three years after baseline, independently of baseline level of symptoms, and other child and family characteristics.

#### **Background**

#### **ADHD**

Attention-Deficit/Hyperactivity Disorder (ADHD) is a neuropsychiatric disorder characterized by disturbances of activity, impulsivity, and attention. It is the most frequent diagnosis in child- and adolescent psychiatry in Denmark (Classified as Hyperkinetic Disorder according to ICD-10¹) and recently a population based Danish study reported a prevalence of approximately 3% in 11-12 year-old children², while the Danish prevalence by DSM-IV diagnostic classification³ was reported to be approximately 6 % in 8-9 year-old children⁴. The estimated worldwide DSM-IV prevalence is approximately 5 % in school children⁵. Recent research suggests that the aetiology of ADHD combines genetic, pre- and perinatal risk factors, and other environmental and psychosocial risk factors, which probably are interrelated in a gene-environment interplay ⁶. The heritability of ADHD is high <sup>7,8</sup>, and the disorder frequently occurs simultaneously in several members of a family <sup>9,10</sup>.

Moreover, according to clinical studies psychiatric comorbidity occurs in 70-80 % of children with ADHD<sup>11,12</sup>, such as sleep disorder, oppositional defiant- or conduct disorder, tic disorders, anxiety- and depressive disorders, and learning and developmental disorders. Recently, a Danish nationwide registry study reported a comorbidity rate of 52% in children and adolescents according to ICD-10 criteria over a sixteen-year period <sup>13</sup>. The lower rate of comorbidity in this registry study could perhaps be explained by the fact that there are daily clinical routine practices and diagnostic traditions in the country.

Long-term studies indicate that ADHD often persists into adulthood<sup>14,15</sup> and is associated with problems in the domains of education, personal relationships, employment status, self-esteem, secondary psychiatric disorders, substance abuse, and criminality<sup>14,16-21</sup>. Successful treatment in childhood may improve child development, daily functioning, school attendance and learning, and thereby potentially also the prognosis and may reduce the societal costs of ADHD<sup>20,22-27</sup>. Thus, there is a strong need, both on the individual and the societal level, to further map out the evidence of factors that moderate the effect and the treatment compliance of children with ADHD.

#### **Treatment**

Psychosocial treatment guided by the symptoms of the child and the needs of the family is mandatory in childhood ADHD. In moderate to severe ADHD, Danish and international guidelines specify the combination of psychosocial treatment and drug treatment with methylphenidate (MPH) as the first line treatment. However, drug treatment is not indicated for all children with ADHD and the indication for continuous treatment needs regular assessment <sup>28-30</sup>.

MPH treatment has a beneficial effect on the core symptoms of ADHD and academic performance in approximately 70% of the children with ADHD <sup>31,32</sup> and a significantly better general function in medicated children with ADHD has been reported<sup>28</sup>. Furthermore, drug treatment may have a protective effect on risk behaviors associated with ADHD, such as accidents, substance abuse, and criminality. A Swedish registry based study assessing criminality rates in adolescents(≥15 years old) and adults diagnosed with ADHD, reported a significant reduction in criminality rates during periods with ADHD medication<sup>33,34</sup>. The long term effects of drug treatment of ADHD are less well studied, but recent data have demonstrated a protective long-term effect on the development of substance abuse <sup>20,35</sup>, suicidal behavior<sup>23</sup>, self-esteem, and social- and academic functioning <sup>26,36</sup>. A Danish registry based study, covering a total of 20.742 patients with ADHD, has recently reported that patients medicated with MPH only, had the lowest rate of substance use disorder<sup>37</sup>.

However, studies on adherence indicate a rather high discontinuation rate of ADHD-medication of 53 % within the first 6-12 months of treatment<sup>38-41</sup>, and up to 80 % after 36 months<sup>42-44</sup>. Early non-compliance has been associated with advanced age of the child, younger parental age, severity of ADHD core symptoms and conduct disorder<sup>38,44</sup>. Parental experience of poor treatment effect, side effects, especially psychological effects such as mood changes and irritability, or the child's reluctance or forgetfulness in relation to medication have been frequently identified as reasons for treatment discontinuation<sup>39,45</sup>.

The Multimodal Treatment Study of Children With Attention-Deficit/Hyperactivity Disorder (MTA)<sup>46</sup> measured saliva MPH concentration at four time points during a 14 months treatment period. Only 53% of the participants were adherent at every time point. In addition, non-adherence resulted in greater deterioration of function in children in the medication-only group, compared to the group receiving both pharmacological and psychosocial treatment<sup>41</sup>. This study emphasized the importance of a psychosocial treatment program in combination with drug treatment.

#### Psychosocial aspects of childhood ADHD

The importance of the psychosocial environment on the effectiveness and compliance in pharmacological treatment of ADHD has only sparsely been described. A recent British study of 570 children with ADHD recruited from child and adolescent psychiatry and pediatric services with a mean age of 10,78 years reported a parental rate of ADHD as high as 29 % <sup>54</sup>. The symptom load in the parents was associated with greater ADHD symptom severity in the child, comorbid Conduct Disorder, higher levels of conflict and lower levels of cohesion in the family.

Likewise, the impact of having a child with ADHD on the parents should not be underestimated. A recent register based Danish study reported a significant negative association between a diagnosis of ADHD in the first born child, and stability of parental relationship and labor market attachment<sup>55</sup>. In addition, ADHD symptoms in the child and behavior seem to evoke maternal hostility, regardless of maternal status of ADHD<sup>56</sup>.

The eight year prospective follow-up study of the MTA cohort concluded that early clinical presentation and function, socio-demographic advantage, and a good initial response to any kind of treatment predicted the best long- term prognosis<sup>57</sup>. A recent Canadian study followed a population-based birth cohort of 1920 children from the age of 5 months to 10 years. Socio-demographic baseline data, children's mental health symptoms, and parenting practices were assessed by questionnaires at baseline and at 6 time points during the follow-up period. The strongest predictor of ADHD medication use, beside ADHD symptoms, was low maternal education, whereas immigrant status lowered the likelihood of medication use<sup>58</sup>. This study relied solely on parental questionnaires and no data of diagnoses, functional impairment and adherence to treatment was obtained.

An increased knowledge of these associations and predictors, based on data from the national Danish registers, could contribute to the development of more differentiated treatment programs. Moreover, it could contribute to the identification of patients and families in need of a more intensive and broadspectrum treatment and monitoring program.

#### Functional impairment

Overall, ADHD has a negative effect on the quality of life of children, which is comparable to severe physical disorders. Recent data suggest that this effect is mediated by an impaired daily functional level in the areas of education and social interaction<sup>59</sup>. The combination of ADHD core symptoms, emotional dysregulation, comorbidity, and learning difficulties causes a marked impairment in behavioral, social, and academic functioning which is beyond what might be expected based on the ADHD core symptoms alone<sup>59,60</sup>. Often families specify the wish to improve the child's academic and social functioning at school and his or her interaction with friends and the family. This is the main reason for seeking treatment of ADHD, rather than ADHD core symptoms alone<sup>61</sup>.

#### **Materials and methods**

#### **Participants**

The design is a longitudinal, naturalistic study of a clinical cohort of 200 drug-naïve children, aged 7-12 years, followed up closely with respect to the beneficial and adverse effects during the first 12 weeks of MPH treatment at the Child and Adolescent Mental Health Center – Capital Region of Denmark<sup>62</sup>. The recruitment was completed in August 2014 and the three months follow-up was completed in November 2014 with patient data recorded in a research database.

#### **Methods**

#### **Recruitment and assessment**

A schematic outline of the assessments over time is given below. We have examined and diagnosed 200 referred children with ADHD based on a clinical assessment, a diagnostic interview (Schedule for affective disorders and schizophrenia for school-aged children(K-SADS-PL)<sup>63</sup>, rating scales (Child Behavior Checklist, CBCL and Teacher Report Form<sup>64-66</sup>, Weiss Functional Impairment Rating Scale-Parent Report, WFIRS-P <sup>67,68</sup>, ADHD-Rating Scale, ADHD-RS <sup>69,70</sup>, and a computerized test of attention and impulsivity (Test of Variables of Attention, TOVA <sup>71</sup>). Children were diagnosed according to both ICD-10 and DSM-IV criteria.

The following rating scales were used both at baseline (t1) and after 3 months (t2) of MPH treatment: Clinician rated ADHD-DSM-IV-RS<sup>72</sup>, Clinical Global Impression (CGI)- Severity <sup>73</sup>, CGI-Improvement, Barkleys Side Effect Rating Scale modified with questions of cardiovascular symptoms, parent and teacher rated ADHD-RS, WFIRS-P, and finally a TOVA test.

At the 36 months (t3) follow-up we will send out the following questionnaires to parents: ADHD-RS, and WFIRS-P

**ADHD core symptoms:** The ADHD core symptom severity was measured by parent- and teacher-rated ADHD-RS, and clinician-rated ADHD-DSM-IV-RS.

**Level of psychosocial functioning:** The level of daily- and social functioning was measured by the WFIRS-P, which is a parent rated questionnaire for assessment of functional impairment within six domains: Academic (learning and behavior), family, life skills, self-perception, social activities, risky activities. The WFIRS-P is a psychometric questionnaire which has been used in several studies for assessment of

treatment related changes in ADHD<sup>74-76</sup>. The psychometric properties of WFIRS-P are investigated in an ongoing project at the Child and Adolescent Mental Health Center – Capital Region of Denmark<sup>77</sup>.

#### Data from the national registers

We will apply for permission to use the following data from several national registers to allow for a thorough analysis of risk and psychosocial factors.

Danish Medical Birth Register: Gestational age, birth weight, Apgar score, birth complications, maternal smoking during pregnancy

Danish Civil Registration System: Age of parents and siblings, ethnicity (parental country of birth)

Integrated Database for Longitudinal Labour Market Research (IDA): Education of mother and father (level and duration), employment status, income, and marital status

Danish National Hospital Register: Lifetime somatic diagnoses of the index child

Danish Psychiatric Central Register: Lifetime psychiatric diagnoses of index child, parents and siblings.

#### Danish Prescription Registry:

ADHD medication prescribed and purchased by the cohort in the 36 months follow-up period, in particular the frequency of dispensed prescriptions (methylphenidate (ATC code N06BA04), dexamfetamine (N06BA02) or atomoxetine (N06BA09)), as well as the date of the first and the last dispensed prescription in the follow-up period. Dosage will be defined as DDD (defined daily dosages) and depending on the distributions duration and dosage will be treated either as continuous or categorical variables in the analyses.

#### **Analyses**

The hypotheses of the study will be tested, with the following data either assessed at baseline, or collected from the national registers, or re-assessed in the follow-up study:

The predictive value of responder status in week three and week 12 for the ADHD-RS score and WFIRS-P score after three years will be tested with ANOVAs. Adjusted R2 will be used as a measure of the proportion of the variation in the outcome variables explained by potential predictors.

To select the best model of predictors for outcome after three years, multiple linear regression analyses will be carried out, with three models of predictors. Model one includes gender, age group (</≥ 10 years), comorbidity (none versus ≥ 1 comorbid diagnosis), IQ (full scale IQ > 85/70-85), maternal education (primary and lower secondary, upper secondary, higher), parental psychiatric disorder (none/ any maternal or parental disorder), baseline ADHD-RS total score. In model two responder status in week three will be added. In model three responder status in week 12 will be added and responder status in week three removed, to test if this is a better model of predictors.

We will perform QQ plots of the outcome variables in the multiple linear regression analyses. Paired-samples T-tests will be used to explore the development and significant changes in impairment in daily life and social functioning as measured by WFIRS-P.

To explore the relation between symptomatology (ADHD-RS) and impairment in daily life and social functioning (WFIRS-P) correlations between scores at baseline, week 12 and year three will be computed.

We will also investigate the moderating effect of pharmacological treatment of ADHD on ADHD symptom score and functional impairment in daily life, after 3 and after 36 months of follow-up in separate studies.

#### Innovative value and perspective of the project

From a clinical perspective, the project will provide new insights and recommendations how to individualize and improve the treatment of children with ADHD. Thus, the project will have an impact on clinical practice and services provided to this clientele.

From a scientific perspective, the project will provide new knowledge about predictors for successful treatment of ADHD, and for the long-term symptomatic and functional outcome in this disorder. The systematic and prospective collection of baseline data, data on symptoms, functional impairment, and treatment effect during the first 3 months of treatment on all children in the cohort, in combination with selected data from the registries is a unique feature of this study. In addition, attrition analyses can be performed to study the impact of baseline and risk factors on dropping out of the study at 36 months follow-up.

In a future perspective, these data combined with data from the 36 months follow-up study might constitute a unique cohort, which can be followed and linked to genetic and other biological data derived from blood samples of the participants. At this time, all participants (or there guardians, respectively) have consented already, to participate in the Gene and Environment Study<sup>78</sup>

#### **Ethical considerations**

The baseline and 3 months follow-up data have already been collected with a protocol that is covered by existing permissions from the local committees on scientific ethics (De Videnskabsetiske Komiteer for Region Hovedstaden) and the Danish Data Protection Agency (Datatilsynet). These permissions allow the collection and examination of data as well as biological specimens from psychiatric patients below the age of 18 years for research purposes. The parents have given informed consent to the data collection. The local committees on scientific ethics in the Capital Region of Denmark and the Danish Data Protection Agency have given permission to collect data from the national registers and the 36-month follow-up study. The latter consists of two parental questionnaires (overall duration about 20 min). The data collected in the study and from the registers will be linked anonymously.

#### Intellectual and scientific environment of the project

The project is conducted by the Research Unit at the Child and Adolescent Mental Health Center, Mental Health Services - Capital Region of Denmark, headed by Professor Anne-Katrine Pagsberg. The principal supervisor is Professor Frank Verhulst. Pia Jeppesen, Ph.D., senior researcher and consultant, and Professor Niels Bilenberg, Department of Child and Adolescent Psychiatry, University of Southern Denmark, Odense, will collaborate and serve as expert consultants on the study.

The project will be carried out by consultant Tine Houmann, head of the unit for preschool-children at the Child and Adolescent Mental Health Center. Collaborators in data collection and analyzes are Kristine K. Jørgensen MD, Ph.D.-student at the Center for Child and Adolescent Mental Health, Mental Health Services, the Capital Region of Denmark; and Henrik Berg Rasmussen, Ph.D, senior researcher at the Institute of Biological Psychiatry, Mental Health Centre Sct. Hans, Mental Health Services, the Capital Region of Denmark.

#### Reference List

- (1) World Health Organisation. The ICD-10 Classification of Mental and Behavioural Disorders, Diagnostic criteria for research. Geneva: 1993.
- (2) Rimvall MK, Elberling H, Rask CU, Helenius D, Skovgaard AM, Jeppesen P. Predicting ADHD in school age when using the Strengths and Difficulties Questionnaire in preschool

age: a longitudinal general population study, CCC2000.

2014

Eur Child Adolesc Psychiatry 2014.

- (3) American Psychiatric Association. Diagnostic and Statistical Manual of mental Disorders-IV. 4 ed. 1994.
- (4) Petersen DJ, Bilenberg N, Hoerder K, Gillberg C.

The population prevalence of child psychiatric disorders in Danish 8- to 9-year-old children.

2006

Eur Child Adolesc Psychiatry 2006;15(2):71-8.

(5) Polanczyk G, Rohde LA.

Epidemiology of attention-deficit/hyperactivity disorder across the lifespan.

2007

Curr Opin Psychiatry 2007;20(4):386-92.

(6) Thapar A, Cooper M, Eyre O, Langley K.

What have we learnt about the causes of ADHD?

2013

J Child Psychol Psychiatry 2013;54(1):3-16.

(7) Nikolas MA, Burt SA.

Genetic and environmental influences on ADHD symptom dimensions of inattention and hyperactivity: a meta-analysis.

2010

J Abnorm Psychol 2010;119(1):1-17.

(8) Faraone SV.

The scientific foundation for understanding attention-deficit/hyperactivity disorder as a valid psychiatric disorder.

2005

Eur Child Adolesc Psychiatry 2005;14(1):1-10.

(9) Agha SS, Zammit S, Thapar A, Langley K.

Are parental ADHD problems associated with a more severe clinical presentation and greater family adversity in children with ADHD?

2013

Eur Child Adolesc Psychiatry 2013;22(6):369-77.

(10) Faraone SV, Biederman J, Mick E, Williamson S, Wilens T, Spencer T, et al.

Family study of girls with attention deficit hyperactivity disorder.

Am J Psychiatry 2000;157(7):1077-83.

(11) Wilens TE, Biederman J, Brown S, Tanguay S, Monuteaux MC, Blake C, et al.

Psychiatric comorbidity and functioning in clinically referred preschool children and school-age youths with ADHD.

2002

J Am Acad Child Adolesc Psychiatry 2002;41(3):262-8.

(12) Kadesjo B, Gillberg C.

The comorbidity of ADHD in the general population of Swedish school-age children.

2001

J Child Psychol Psychiatry 2001;42(4):487-92.

(13) Jensen CM, Steinhausen HC.

Comorbid mental disorders in children and adolescents with attention-deficit/hyperactivity disorder in a large nationwide study.

2014

Atten Defic Hyperact Disord 2014.

(14) Biederman J, Petty CR, Woodworth KY, Lomedico A, Hyder LL, Faraone SV.

Adult outcome of attention-deficit/hyperactivity disorder: a controlled 16-year follow-up study. 2012

J Clin Psychiatry 2012;73(7):941-50.

(15) Faraone SV, Biederman J, Mick E.

The age-dependent decline of attention deficit hyperactivity disorder: a meta-analysis of follow-up studies.

2006

Psychol Med 2006;36(2):159-65.

(16) Langley K, Fowler T, Ford T, Thapar AK, van den BM, Harold G, et al.

Adolescent clinical outcomes for young people with attention-deficit hyperactivity disorder. 2010

Br J Psychiatry 2010;196(3):235-40.

(17) Hinshaw SP, Owens EB, Sami N, Fargeon S.

Prospective follow-up of girls with attention-deficit/hyperactivity disorder into adolescence: Evidence for continuing cross-domain impairment.

2006

J Consult Clin Psychol 2006;74(3):489-99.

(18) Hinshaw SP, Owens EB, Zalecki C, Huggins SP, Montenegro-Nevado AJ, Schrodek E, et al.

Prospective follow-up of girls with attention-deficit/hyperactivity disorder into early adulthood: continuing impairment includes elevated risk for suicide attempts and self-injury. 2012

J Consult Clin Psychol 2012;80(6):1041-51.

(19) Dalsgaard S, Mortensen PB, Frydenberg M, Thomsen PH.

Long-term criminal outcome of children with attention deficit hyperactivity disorder.

Crim Behav Ment Health 2013;23(2):86-98.

(20) Dalsgaard S, Mortensen PB, Frydenberg M, Thomsen PH.

ADHD, stimulant treatment in childhood and subsequent substance abuse in adulthood - a naturalistic long-term follow-up study.

2014

Addict Behav 2014;39(1):325-8.

(21) Dalsgaard S, Mortensen PB, Frydenberg M, Thomsen PH.

Conduct problems, gender and adult psychiatric outcome of children with attention-deficit hyperactivity disorder.

2002

Br J Psychiatry 2002;181:416-21.

(22) Dalsgaard S, Nielsen HS, Simonsen M.

Consequences of ADHD medication use for children's outcomes.

2014

J Health Econ 2014;37:137-51.

(23) Chen Q, Sjolander A, Runeson B, D'Onofrio BM, Lichtenstein P, Larsson H.

Drug treatment for attention-deficit/hyperactivity disorder and suicidal behaviour: register based study.

2014

BMJ 2014;348:g3769.

(24) Holden SE, Jenkins-Jones S, Poole CD, Morgan CL, Coghill D, Currie CJ.

The prevalence and incidence, resource use and financial costs of treating people with attention deficit/hyperactivity disorder (ADHD) in the United Kingdom (1998 to 2010).

2013

Child Adolesc Psychiatry Ment Health 2013;7(1):34.

(25) Coghill D, Soutullo C, d'Aubuisson C, Preuss U, Lindback T, Silverberg M, et al.

Impact of attention-deficit/hyperactivity disorder on the patient and family: results from a European survey.

2008

Child Adolesc Psychiatry Ment Health 2008;2(1):31.

(26) Shaw M, Hodgkins P, Caci H, Young S, Kahle J, Woods AG, et al.

A systematic review and analysis of long-term outcomes in attention deficit hyperactivity disorder: effects of treatment and non-treatment.

2012

BMC Med 2012;10:99.

(27) Le HH, Hodgkins P, Postma MJ, Kahle J, Sikirica V, Setyawan J, et al.

Economic impact of childhood/adolescent ADHD in a European setting: the Netherlands as a reference case.

2014

Eur Child Adolesc Psychiatry 2014;23(7):587-98.

- (28) National Institute for Health and Clinical Excellence. Attention deficit hyperactivity disorder. Nice clinical guideline 72 2008Available from: URL: www.nice.org.uk/CG072
- (29) Sundhedsstyrelsen. National klinisk retningslinje for udredning og behandling af ADHD hos børn og unge. <a href="http://sundhedsstyrelsen">http://sundhedsstyrelsen</a>

dk/da/nyheder/2014/~/media/A7931B11333540A184C73465181E29CE ashx 2014 [cited 2014 May 23];Available from: URL: <a href="http://sst.dk">http://sst.dk</a>

(30) Pliszka S.

Practice parameter for the assessment and treatment of children and adolescents with attention-deficit/hyperactivity disorder.

2007

J Am Acad Child Adolesc Psychiatry 2007;46(7):894-921.

(31) Banaschewski T, Coghill D, Santosh P, Zuddas A, Asherson P, Buitelaar J, et al.

Long-acting medications for the hyperkinetic disorders. A systematic review and European treatment guideline.

2006

Eur Child Adolesc Psychiatry 2006;15(8):476-95.

(32) Prasad V, Brogan E, Mulvaney C, Grainge M, Stanton W, Sayal K.

How effective are drug treatments for children with ADHD at improving on-task behaviour and academic achievement in the school classroom? A systematic review and meta-analysis. 2013

Eur Child Adolesc Psychiatry 2013;22(4):203-16.

(33) van de Loo-Neus GH, Rommelse N, Buitelaar JK.

To stop or not to stop? How long should medication treatment of attention-deficit hyperactivity disorder be extended?

2011

Eur Neuropsychopharmacol 2011;21(8):584-99.

(34) Lichtenstein P, Halldner L, Zetterqvist J, Sjolander A, Serlachius E, Fazel S, et al.

Medication for attention deficit-hyperactivity disorder and criminality.

2012

N Engl J Med 2012;367(21):2006-14.

(35) Groenman AP, Oosterlaan J, Rommelse NN, Franke B, Greven CU, Hoekstra PJ, et al.

Stimulant treatment for attention-deficit hyperactivity disorder and risk of developing substance use disorder.

2013

Br J Psychiatry 2013;203(2):112-9.

(36) Harpin V, Mazzone L, Raynaud JP, Kahle J, Hodgkins P.

Long-Term Outcomes of ADHD: A Systematic Review of Self-Esteem and Social Function. 2013

J Atten Disord 2013.

(37) Steinhausen HC, Bisgaard C.

Substance use disorders in association with attention-deficit/hyperactivity disorder, co-morbid mental disorders, and medication in a nationwide sample.

Eur Neuropsychopharmacol 2014;24(2):232-41.

(38) Hong M, Lee WH, Moon DS, Lee SM, Chung US, Bahn GH.

A 36 month naturalistic retrospective study of clinic-treated youth with attention-deficit/hyperactivity disorder.

2014

J Child Adolesc Psychopharmacol 2014;24(6):341-6.

(39) Toomey SL, Sox CM, Rusinak D, Finkelstein JA.

Why do children with ADHD discontinue their medication?

2012

Clin Pediatr (Phila) 2012;51(8):763-9.

(40) Garbe E, Mikolajczyk RT, Banaschewski T, Petermann U, Petermann F, Kraut AA, et al.

Drug treatment patterns of attention-deficit/hyperactivity disorder in children and adolescents in Germany: results from a large population-based cohort study.

2012

J Child Adolesc Psychopharmacol 2012;22(6):452-8.

(41) Pappadopulos E, Jensen PS, Chait AR, Arnold LE, Swanson JM, Greenhill LL, et al.

Medication adherence in the MTA: saliva methylphenidate samples versus parent report and mediating effect of concomitant behavioral treatment.

2009

J Am Acad Child Adolesc Psychiatry 2009;48(5):501-10.

(42) Charach A, Gajaria A.

Improving psychostimulant adherence in children with ADHD.

2008

Expert Rev Neurother 2008;8(10):1563-71.

(43) Pottegard A, Bjerregaard BK, Glintborg D, Kortegaard LS, Hallas J, Moreno SI.

The use of medication against attention deficit/hyperactivity disorder in Denmark: a drug use study from a patient perspective.

2013

Eur J Clin Pharmacol 2013;69(3):589-98.

(44) Thiruchelvam D, Charach A, Schachar RJ.

Moderators and mediators of long-term adherence to stimulant treatment in children with ADHD. 2001

J Am Acad Child Adolesc Psychiatry 2001;40(8):922-8.

(45) Gau SS, Shen HY, Chou MC, Tang CS, Chiu YN, Gau CS.

Determinants of adherence to methylphenidate and the impact of poor adherence on maternal and family measures.

2006

J Child Adolesc Psychopharmacol 2006;16(3):286-97.

(46) The MTA Cooperative Group.

A 14-month randomized clinical trial of treatment strategies for attention-deficit/hyperactivity disorder. The MTA Cooperative Group. Multimodal Treatment Study of Children with ADHD.

Arch Gen Psychiatry 1999;56(12):1073-86.

(47) Sobanski E, Banaschewski T, Asherson P, Buitelaar J, Chen W, Franke B, et al.

Emotional lability in children and adolescents with attention deficit/hyperactivity disorder (ADHD): clinical correlates and familial prevalence.

2010

J Child Psychol Psychiatry 2010;51(8):915-23.

(48) Stringaris A, Goodman R.

Mood lability and psychopathology in youth.

2009

Psychol Med 2009;39(8):1237-45.

(49) Shaw P, Stringaris A, Nigg J, Leibenluft E.

Emotion dysregulation in attention deficit hyperactivity disorder.

2014

Am J Psychiatry 2014;171(3):276-93.

(50) Biederman J, Petty CR, Day H, Goldin RL, Spencer T, Faraone SV, et al.

Severity of the aggression/anxiety-depression/attention child behavior checklist profile discriminates between different levels of deficits in emotional regulation in youth with attention-deficit hyperactivity disorder.

2012

J Dev Behav Pediatr 2012;33(3):236-43.

(51) Spencer TJ, Faraone SV, Surman CB, Petty C, Clarke A, Batchelder H, et al.

Toward defining deficient emotional self-regulation in children with attention-deficit/hyperactivity disorder using the Child Behavior Checklist: a controlled study.

2011

Postgrad Med 2011;123(5):50-9.

(52) Kim J, Carlson GA, Meyer SE, Bufferd SJ, Dougherty LR, Dyson MW, et al.

Correlates of the CBCL-dysregulation profile in preschool-aged children.

2012

J Child Psychol Psychiatry 2012;53(9):918-26.

(53) Althoff RR, Verhulst FC, Rettew DC, Hudziak JJ, van der EJ.

Adult outcomes of childhood dysregulation: a 14-year follow-up study.

2010

J Am Acad Child Adolesc Psychiatry 2010;49(11):1105-16.

(54) Agha SS, Zammit S, Thapar A, Langley K.

Are parental ADHD problems associated with a more severe clinical presentation and greater family adversity in children with ADHD?

2013

Eur Child Adolesc Psychiatry 2013;22(6):369-77.

(55) Kvist AP, Nielsen HS, Simonsen M.

The importance of children's ADHD for parents' relationship stability and labor supply.

Soc Sci Med 2013;88:30-8.

(56) Harold GT, Leve LD, Barrett D, Elam K, Neiderhiser JM, Natsuaki MN, et al.

Biological and rearing mother influences on child ADHD symptoms: revisiting the developmental interface between nature and nurture.

2013

J Child Psychol Psychiatry 2013;54(10):1038-46.

(57) Molina BS, Hinshaw SP, Swanson JM, Arnold LE, Vitiello B, Jensen PS, et al.

The MTA at 8 years: prospective follow-up of children treated for combined-type ADHD in a multisite study.

2009

J Am Acad Child Adolesc Psychiatry 2009;48(5):484-500.

(58) Galera C, Pingault JB, Michel G, Bouvard MP, Melchior M, Falissard B, et al.

Clinical and social factors associated with attention-deficit hyperactivity disorder medication use: population-based longitudinal study.

2014

Br J Psychiatry 2014;205(4):291-7.

(59) Danckaerts M, Sonuga-Barke EJ, Banaschewski T, Buitelaar J, Dopfner M, Hollis C, et al.

The quality of life of children with attention deficit/hyperactivity disorder: a systematic review. 2010

Eur Child Adolesc Psychiatry 2010;19(2):83-105.

(60) Coghill D, Danckaerts M, Sonuga-Barke E, Sergeant J.

Practitioner review: Quality of life in child mental health--conceptual challenges and practical choices.

2009

J Child Psychol Psychiatry 2009;50(5):544-61.

(61) Parens E, Johnston J.

Facts, values, and attention-deficit hyperactivity disorder (ADHD): an update on the controversies. 2009

Child Adolesc Psychiatry Ment Health 2009;3(1):1.

- (62) INDICES-WP6. <a href="http://forskning">http://forskning</a> regionh dk/psykiatrien/da/projects/sammenhaengen-mellem-ces1-genotype-og-methylphenidat-respons-hos-boern-med-adhd-indices-arbejdspakke-6--et-phdstudie(bdea93e8-e711-4742-a28a-06d9e1e2f20d) html 2014Available from: URL: <a href="http://forskning.regionh.dk/psykiatrien/da/projects/sammenhaengen-mellem-ces1-genotype-og-methylphenidat-respons-hos-boern-med-adhd-indices-arbejdspakke-6--et-phdstudie(bdea93e8-e711-4742-a28a-06d9e1e2f20d).html</a>
- (63) Ambrosini PJ.

Historical development and present status of the schedule for affective disorders and schizophrenia for school-age children (K-SADS).

2000

J Am Acad Child Adolesc Psychiatry 2000;39(1):49-58.

(64) Achenbach T.M. Manual for the child Behavior Checklist/4-18 and 1991 Profile. Burlington VT: University of Vermont Department of Psychiatry; 1991.

#### (65) Bilenberg N.

The Child Behavior Checklist (CBCL) and related material: standardization and validation in Danish population based and clinically based samples.

1999

Acta Psychiatr Scand Suppl 1999;398:2-52.

(66) Henriksen J, Nielsen PF, Bilenberg N.

New Danish standardization of the Child Behaviour Checklist.

2012

Dan Med J 2012;59(7):A4462.

(67) Epstein JN, Weiss MD.

Assessing treatment outcomes in attention-deficit/hyperactivity disorder: a narrative review. 2012

Prim Care Companion CNS Disord 2012;14(6).

- (68) Clinical Trials WFIRS. <a href="http://clinicaltrialsfeeds">http://clinicaltrialsfeeds</a> org/clinical-trials/results/term=WFIRS 2013Available from: URL: <a href="http://clinicaltrialsfeeds.org/clinical-trials/results/term=WFIRS">http://clinicaltrialsfeeds.org/clinical-trials/results/term=WFIRS</a>.
- (69) Barkley RA, Gwenyth EH, Arthur LR. Defiant Teens. A Clinician's Manual for Assessment and Family Intervention. New York: The Guilford Press; 1999.
- (70) Szomlaiski N, Dyrborg J, Rasmussen H, Schumann T, Koch SV, Bilenberg N.
  Validity and clinical feasibility of the ADHD rating scale (ADHD-RS) A Danish Nationwide Multicenter Study.

2009

Acta Paediatr 2009;98(2):397-402.

(71) Schatz AM, Ballantyne AO, Trauner DA.

Sensitivity and specificity of a computerized test of attention in the diagnosis of Attention-Deficit/Hyperactivity Disorder.

2001

Assessment 2001;8(4):357-65.

- (72) DuPaul GJ, Power TJ, Anastopoulos A, Reid R. ADHD Rating Scale IV. New York: The Guilford Press; 1998.
- (73) Berk M, Ng F, Dodd S, Callaly T, Campbell S, Bernardo M, et al.

The validity of the CGI severity and improvement scales as measures of clinical effectiveness suitable for routine clinical use.

2008

J Eval Clin Pract 2008;14(6):979-83.

(74) Banaschewski T, Soutullo C, Lecendreux M, Johnson M, Zuddas A, Hodgkins P, et al. Health-related quality of life and functional outcomes from a randomized, controlled study of lisdexamfetamine dimesylate in children and adolescents with attention deficit hyperactivity disorder. 2013 CNS Drugs 2013;27(10):829-40.

(75) Stein MA, Waldman ID, Charney E, Aryal S, Sable C, Gruber R, et al. Dose effects and comparative effectiveness of extended release dexmethylphenidate and mixed amphetamine salts. 2011

J Child Adolesc Psychopharmacol 2011;21(6):581-8.

(76) Hantson J, Wang PP, Grizenko-Vida M, Ter-Stepanian M, Harvey W, Joober R, et al.
 Effectiveness of a therapeutic summer camp for children with ADHD: Phase I Clinical Intervention Trial.
 2012
 J Atten Disord 2012;16(7):610-7.

- (77) Vurdering af det daglige funktionsniveau hos børn med ADHD en undersøgelse af funktionsskalaen WFIRS. <a href="http://forskning">http://forskning</a> regionh dk/psykiatrien/da/projects/vurdering-af-det-daglige-funktionsniveau-hos-boern-med-adhd--en-undersoegelse-af-funktionsskalaen-wfirs(c52b1465-34a7-4231-a15e-10d12f631ba7) html 2014Available from: URL: <a href="http://forskning.regionh.dk/psykiatrien/da/projects/vurdering-af-det-daglige-funktionsniveau-hos-boern-med-adhd--en-undersoegelse-af-funktionsskalaen-wfirs(c52b1465-34a7-4231-a15e-10d12f631ba7).html</p>
- (78) Pagsberg AK, Werge T.M. Arv og Miljø. <a href="http://forskning">http://forskning</a> regionh dk/psykiatrien/da/projects/arv-og-miljoe(18fa29b1-80fa-4b87-837e-a0215f1bfc8f) html 2015Available from: URL: <a href="http://forskning.regionh.dk/psykiatrien/da/projects/arv-og-miljoe(18fa29b1-80fa-4b87-837e-a0215f1bfc8f]">http://forskning.regionh.dk/psykiatrien/da/projects/arv-og-miljoe(18fa29b1-80fa-4b87-837e-a0215f1bfc8f]</a>).html

### Summary of amendments to study protocol

| Protocol version | Date of approval | Revisions |
|---|---|---|
| Original protocol | Approval from human subject protection review board: 22 <sup>nd</sup> March 2012 | Original version approved by the local scientific ethics committee (Journal nr.:H-B-2009-026) |
| Additional protocol | Approval from human subject protection review board: N/A | The additional protocol includes questionnaires and retrospective data extraction from registers and patient journals. |
| | Latest approval for data extraction: 22 <sup>nd</sup> November 2016 | The local scientific ethics committee deemed this addition not applicable for ethical review. |